CLINICAL TRIAL: NCT04227704
Title: Postpartum Depression After Cesarean Delivery: Ketamine as a Preventative Intervention: A Feasibility Pilot-study
Brief Title: Ketamine to Prevent PPD After Cesarean
Acronym: PoCKet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, David Monks, Asst Prof of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201910191
Record Dates: First submitted 2019-11-20; First posted 2020-01-14 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of three groups (two interventional and one control).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The ketamine and placebo study injectates (subcutaneous and intravenous) will be prepared, in way that does not allow differentiation, by pharmacy staff who are otherwise uninvolved in the study. Participants will be allocated to groups using a random sequence generator. The patients, investigators and outcome assessors will remain unaware of their group until data collection is complete for all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Shortly after cesarean delivery of their baby, participants will receive a subcutaneous injection and 40-minute intravenous infusion of 0.9% sodium chloride.
  Interventions: Drug: Control
- Ketamine SC (Experimental): Shortly after cesarean delivery of their baby, participants will receive a subcutaneous injection of 0.5 mg/kg of ketamine and a 40-minute intravenous infusion of 0.9% sodium chloride.
  Interventions: Drug: Ketamine 50 MG/ML; Drug: Control
- Ketamine IVI (Experimental): Shortly after cesarean delivery of their baby, participants will receive a subcutaneous injection of 0.9% sodium chloride and a 40-minute intravenous infusion of 0.5 mg/kg ketamine.
  Interventions: Drug: Ketamine 50 MG/ML; Drug: Control

INTERVENTIONS:
Drug: Ketamine 50 MG/ML — Administration of a 0.5 mg/kg dose of ketamine at cesarean delivery by one of two routes (subcutaneous or 40-minute IV infusion).
  Arms: Ketamine IVI; Ketamine SC
Drug: Control — Administration of 0.9% Sodium Chloride (N/S)

SUMMARY:
The investigators plan to randomise participants to receive ketamine or placebo control subcutaneously or by 40-minute intravenous infusions and will follow them up for 42 days to assess the incidence of postpartum depression. This feasibility pilot study is designed to explore the adequacy of the study procedures and tolerability of the interventions.

DETAILED DESCRIPTION:
Postpartum depression (PPD)

PPD is one of the most common perinatal medical complications and can have a detrimental effect on both mother and baby. Suicide exceeds hemorrhage and hypertensive disorders as a cause of maternal mortality and maternal psychopathology interferes with the parent-infant relationship. It has been estimated to have a period prevalence of 19.2% in the first 3 postpartum months. The rapid decline in reproductive hormones is thought to contribute to the development of PPD in susceptible women, although the specific pathogenesis is unknown. The American College of Obstetricians and Gynecologists recommend that all women should be routinely screened for depressive symptoms in the perinatal period.

Risk factors for PPD include:

* Depression during pregnancy • Breastfeeding problems
* Preterm birth/infant admission to neonatal intensive care (NICU)
* Traumatic birth experience
* History of depression
* Anxiety during pregnancy

Ketamine's anti-depressant effect

Ketamine, a phencyclidine derivative, is a non-competitive antagonist at the N-methyl-D-aspartic acid (NMDA) receptor that is commonly used as an anesthetic or sedative agent and has proven analgesic effect after a variety of surgeries including CD, where it has also been shown to reduce shivering. It has been demonstrated to have a rapid anti-depressant effect in treatment-resistant depression outside of pregnancy. The most commonly employed intravenous (IV) dose for this purpose is 0.5 mg/kg over 40 minutes, as single or repeated infusions. It has been postulated that prolonged blockade of NMDA receptors causes long-term changes in signal transduction leading to sustained clinical improvement, some investigators have explored longer term infusions such as those used to treat chronic pain. A recent pilot study assessing the feasibility of a 96-hour (~0.5mg/kg/hr) infusion compared with a single 40-minute (0.5 mg/kg) infusion suggested a trend toward greater efficacy in the prolonged infusion but confirmation of a statistically significant result is awaited.

Ketamine and PPD

This promising anti-depressant effect has prompted investigation of ketamine as a preventative measure in patients undergoing CD. There have been 2 studies to date, one which failed to demonstrate any benefit from a bolus dose of 0.25 mg/kg and one which documented a large reduction (1 and 22% in the treatment and control, respectively) in the (6 week) period prevalence of postpartum depression after a 4 mg/kg dose of ketamine over 50 hours (~0.08 mg/kg/hr).

The prolonged IV infusion, was achieved by adding the ketamine to a sufentanil patient-controlled analgesic (PCA) pump with a background infusion. This PCA pump is a standard part of their post-cesarean analgesic regimen. In our institution, it is standard practice to discontinue IV infusions and to remove IV cannulae as early as it is safe to do so. This practice is essential to the attempts to enhance postoperative recovery and aid mother's bonding with their babies and facilitate their early-life care. This reflects patients' expectations and preferences and is in line with other maternity units across North America and Europe.

The natural course of PPD varies and, although it may resolve spontaneously within weeks, approximately 20% of women with PPD still have depression at 12 months and beyond. As many as 13% will still have depressive symptoms at 2 years and 40% will have a relapse. Considering the maternal suffering, disruption to the family, potential impairment of the social, emotional, and cognitive development of the child, and the rare cases of infanticide and suicide caused by PPD, the impact on families and society as a whole is difficult to overemphasize. An intervention that promises such a large reduction in this devastating disease warrants extensive research. In an attempt to achieve the benefit whilst employing methods more acceptable to our patients we have designed a pilot study to assess the feasibility of our study design and collect preliminary tolerability and efficacy data on ketamine administered by two alternative routes: 40-minute IV infusion (i.v.) and subcutaneous (s.c.) injection.

ELIGIBILITY:
Inclusion criteria:

* Term pregnancy
* Age 18-45 years of age
* Scheduled cesarean delivery under neuraxial anesthesia

Exclusion criteria:

* ASA classification IV or V
* History of psychotic episodes
* History of allergy to ketamine
* Inability to communicate in English or any other barrier to providing informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monks DT, Palanisamy A, Jaffer D, Singh PM, Carter E, Lenze S. A randomized feasibility pilot-study of intravenous and subcutaneous administration of ketamine to prevent postpartum depression after planned cesarean delivery under neuraxial anesthesia. BMC Pregnancy Childbirth. 2022 Oct 21;22(1):786. doi: 10.1186/s12884-022-05118-8. PMID 36271352

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants withdrew from the study; only 23 had data to report.
Period: Overall Study
Arm/Group | Control | Ketamine SC | Ketamine IVI
Started | 8 | 9 | 8
Completed | 7 | 8 | 8
Not Completed | 1 | 1 | 0
Not completed — due to anesthesia being changed to general anesthesia | 0 | 1 | 0
Not completed — due to C/S being cancelled | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketamine SC | Ketamine IVI | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.53) | 32.6 (0.95) | 30.1 (4.30) | 31.8 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 23
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 6 | 5 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 8 | 23
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (7.84) | 41.1 (12.0) | 36.0 (6.06) | 36.8 (9.30)
Gestational age (weeks) [Mean (Standard Deviation); unit: weeks] | 37.5 (.76) | 38.7 (1.11) | 38.0 (1.11) | 38.1 (1.08)
American Society of Anesthesiologists' (ASA) physical status classification system [Count of Participants; unit: Participants] — The purpose of the ASA classification system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning), it can be helpful in predicting perioperative risks. Classified as I - IV, with healthier patients being scored as I and sicker patients as IV.
  Participants
    ASA II | 6 | 5 | 7 | 18
    ASA III | 1 | 3 | 1 | 5
Insurance status [Count of Participants; unit: Participants]
  Insured | 4 | 5 | 6 | 15
  Uninsured | 3 | 3 | 2 | 8
Pre-operative Anxiety, Depression and Psychosocial Stress screening [Mean (Standard Deviation); unit: units on a scale] — General Anxiety Disorder 7-item Scale (GAD-7), ranges from 0 to 21. Higher scores indicate more severe anxiety.
  Edinburgh Postpartum Depression Scale (EPDS) is a set of ten questions assessing mood in the previous seven days. Scored 0-30. Higher scores indicate greater depressive symptomatology.
  The Antenatal Risk Questionnaire (ANRQ) is a patient-reported psychosocial assessment instrument. Scored 0-23, with higher scores indicating higher psychosocial risk factors.
  units on a scale
    Anxiety (GAD-7) | 7.29 (2.93) | 6.13 (8.20) | 6.25 (5.55) | 6.52 (5.81)
    Depression (EPDS) | 8.29 (4.72) | 6.25 (6.27) | 5 (4.78) | 6.43 (5.26)
    Psychosocial stress (ANRQ) | 26.3 (13.0) | 17 (14.4) | 14.9 (9.25) | 19.1 (12.8)
Psychiatric history [Count of Participants; unit: Participants]
  Any psychiatric history | 7 | 2 | 1 | 10
  PPD | 2 | 2 | 0 | 4
  MDD | 3 | 1 | 0 | 4
  Anxiety | 6 | 2 | 2 | 10
  Mood disorder | 2 | 0 | 0 | 2
  Personality disorder | 0 | 0 | 0 | 0
  Psychotic disorder | 0 | 0 | 0 | 0
  Premenstrual syndrome | 0 | 0 | 0 | 0
  Premenstrual dysmorphic disorder | 0 | 0 | 0 | 0
  Panic disorder | 0 | 0 | 1 | 1
  Bipolar affective disorder | 1 | 0 | 0 | 1
  Obsessive compulsive disorder | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of Postpartum Depression in the Study Population, as Defined as EPDS Greater Than 10 Out of 30
Description: Establish a sufficient burden of disease (>10%) in our population to warrant a full RCT
Time Frame: 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 4 | 2 | 5

2. Primary Outcome: Percentage of Eligible Patients Consenting to Participation
Description: Establish a recruitment rate of greater than 50% to confirm the feasibility of conducting an RCT in our population
  Twenty-five (20.7%) out of 121 women who were approached consented to participation. 2 were withdrawn with 23 completing participation.
Time Frame: Through study completion, approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 7 | 8 | 8

3. Primary Outcome: Percentage of Patients With a Complete Dataset
Description: Ensure that the design of assessments and data collection make it possible to achieve a complete dataset in >90% of participants
Time Frame: Through study completion, approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 3 | 4 | 7

4. Primary Outcome: Number of Patients in Study Arms Experiencing One or More Severe Side Effects
Description: Ascertain that neither of the chosen routes of administration of ketamine are intolerable to patients, as defined as the incidence of one or more severe side effects experienced by >10% of participants in that study arm.
Time Frame: Through study completion, approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 0 | 0 | 0

5. Secondary Outcome: Dose of Opiate Analgesics Administered
Description: Intraoperative supplementary analgesia in morphine milligram equivalents
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Morphine Milligram Equivalents | 88.6 (35.6) | 68.4 (63.7) | 67.0 (22.4)

6. Secondary Outcome: Dose of Ketorolac Administered (mg)
Description: Intraoperative supplementary analgesia
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
mg | 30 (0) | 30 (0) | 30 (0)

7. Secondary Outcome: Prevalence of Intraoperative Hypotension
Description: Prevalence of participants with intraoperative hypotension of a systolic BP of less than 90
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 1 | 2 | 1

8. Secondary Outcome: Maximum Intraoperative Pain (NRS)
Description: Reported maximal level of intraoperative pain on the numerical rating scale 0 - 10, where 0 is no pain and 10 is the worst pain imaginable
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Mean (Full Range); unit: Rating Score
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Rating Score | 3 [1 to 5] | 5 [1 to 10] | 1.5 [1 to 5]

9. Secondary Outcome: Adverse Effects
Description: Incidence and severity (mild, moderate or severe) of nausea, vomiting, pruritus, dizziness, sedation, shivering, anxiety, euphoria, hallucinations, amnesia, blurred vision, diplopia, nystagmus
Time Frame: Intraoperative and 2 and 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants
  Mild Nausea | 0 | 2 | 1
  Moderate Nausea | 2 | 0 | 3
  Severe Nausea | 0 | 0 | 0
  Mild vomiting | 0 | 2 | 0
  Moderate vomiting | 1 | 1 | 1
  Severe vomiting | 0 | 0 | 0
  Mild shivering | 6 | 1 | 0
  Moderate shivering | 0 | 1 | 0
  Severe Shivering | 0 | 0 | 0
  Mild sedation | 1 | 1 | 2
  Moderate sedation | 2 | 0 | 1
  Severe sedation | 0 | 0 | 0
  Mild blurred vision | 1 | 1 | 3
  Moderate blurred vision | 0 | 0 | 0
  Severe blurred vision | 0 | 0 | 0
  Mild diplopia | 1 | 0 | 1
  Moderate diplopia | 0 | 0 | 0
  Severe diplopia | 0 | 0 | 0
  Mild dizziness | 1 | 1 | 3
  Moderate dizziness | 0 | 0 | 0
  Severe dizziness | 0 | 0 | 0
  Mild anxiety | 2 | 0 | 1
  Moderate anxiety | 1 | 0 | 0
  Severe anxiety | 0 | 0 | 0
  Mild pruritus | 1 | 4 | 0
  Moderate pruritus | 1 | 0 | 2
  Severe pruritus | 0 | 0 | 0
  Euphoria | 0 | 0 | 0
  Amnesia | 0 | 0 | 0
  Hallucinations | 0 | 0 | 0
  Nystagmus | 0 | 0 | 0

10. Secondary Outcome: Plasma Concentrations of Ketamine
Description: Assays of venous blood samples
Time Frame: At baseline and approximately 20, 40 and 100 minutes postpartum
Population: Ketamine assays not performed and therefore no data collected
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Total Opiate Consumption in Morphine Equivalents
Description: Morphine equivalents
Time Frame: In the first 2 days postpartum
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Morphine Milligram Equivalents | 88.6 (35.6) | 68.4 (63.7) | 67 (22.4)

12. Secondary Outcome: Surgical Site Pain: Numerical Rating Scale (NRS 0-10)
Description: Surgical site pain on a numerical rating scale of 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: At 2, 6, 24 and 48 hours after delivery and on postpartum days 21 and 42
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
units on a scale
  2 hours postoperatively | 2.86 [0 to 9] | 2.1428571428571 [0 to 8] | 2.5 [0 to 6]
  6 hours postoperatively | 3 [0 to 7] | 4.714285714 [2 to 7] | 1.875 [0 to 4]
  24 hours postoperatively | 3 [0 to 7] | 4.571428571 [0 to 9] | 2 [0 to 3]
  48 hours postoperatively | 3.428571429 [0 to 7] | 4.25 [1 to 8] | 3.125 [0 to 7]
  21 days postoperatively | 1 [0 to 3] | 3.333333333 [0 to 8] | 0.875 [0 to 3]
  42 days postoperatively | 0.6666666667 [0 to 2] | 0.333333333 [0 to 2] | 0.285714286 [0 to 1]
Statistical Analysis 1: Comparison: Control vs Ketamine SC vs Ketamine IVI; Test type: Superiority; p = 0.09, ANOVA

13. Secondary Outcome: Edinburgh Postpartum Depression Scale (EPDS)
Description: The EPDS is a validated measure of depressive symptoms in the postpartum period. The scale is scored between 0 - 30, a higher score represents greater depressive symptomatology. We report the study mean of each participant's mean EPDS score for their postpartum assessments
Time Frame: On postpartum days 1, 2, 21 and 42
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
units on a scale
  Day 1 | 7.5 [0 to 13] | 4.75 [0 to 18] | 4.25 [1 to 12]
  Day 2 | 8.43 [0 to 17] | 5.63 [0 to 20] | 5.38 [0 to 12]
  Day 21 | 6.4 [0 to 13] | 2.83 [0 to 8] | 5.14 [0 to 20]
  Day 42 | 9.75 [7 to 17] | 3.33 [0 to 16] | 3.86 [0 to 12]
Statistical Analysis 1: Comparison: Control vs Ketamine SC vs Ketamine IVI; Test type: Superiority; p = 0.08, ANOVA

14. Secondary Outcome: Apgar Scores
Description: Apgar score (0-10) comprised of an assessment of neonatal color, tone and crying. A higher score indicates healthier color, tone and crying.
Time Frame: At 1 and 5 minutes after delivery
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
score on a scale
  Apgar 1min | 8 (1.62) | 8 (2.39) | 8 (0.35)
  Apgar 5 min | 9 (1.83) | 9 (1.16) | 9 (0.46)

15. Secondary Outcome: Admission to NICU
Description: Incidence of admission
Time Frame: Postpartum day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 3 | 1 | 3

16. Secondary Outcome: The Number of Participants Achieving Breastfeeding Success
Description: An indication of whether breastfeeding has been successfully established (Yes or No).
Time Frame: Postpartum days 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants
  Day 1 | 3 | 6 | 5
  Day 2 | 3 | 6 | 5

17. Secondary Outcome: Prevalence of Intraoperative Hypertension
Description: Prevalence of intraoperative hypertension as defined by number of participants with a systolic blood pressure greater than 140 mmHg
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 1 | 0 | 1

18. Secondary Outcome: Prevalence of Intraoperative Bradycardia
Description: Prevalence of intraoperative bradycardia, defined as number of participants with a heart rate of less than 40 bpm
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 0 | 0 | 2

19. Secondary Outcome: Prevalence of Intraoperative Tachycardia
Description: Prevalence of intraoperative tachycardia as defined by the number of participants with a heart rate greater than 110 bpm
Time Frame: Intraoperative phase, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
Participants | 0 | 1 | 1

20. Secondary Outcome: Postpartum Anxiety
Description: Mean Anxiety in the postpartum. General Anxiety Disorder 7-item Scale (GAD-7), ranges from 0 to 21. Higher scores indicate more severe anxiety.
Time Frame: On day of surgery, and postpartum days 1, 2, 21 and 42
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Ketamine SC | Ketamine IVI
Number analyzed (Participants) | 7 | 8 | 8
units on a scale
  Day 1 | 5.17 [0 to 8] | 5.63 [0 to 21] | 3.5 [0 to 12]
  Day 2 | 6 [0 to 13] | 4.75 [0 to 21] | 4.5 [0 to 15]
  Day 21 | 5.8 [0 to 10] | 2.333333333 [0 to 9] | 4.57 [0 to 19]
  Day 42 | 5.75 [4 to 7] | 3.5 [0 to 17] | 2.71 [0 to 9]
Statistical Analysis 1: Comparison: Control vs Ketamine SC vs Ketamine IVI; Test type: Superiority; p = 0.44, ANOVA

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Control | Ketamine SC | Ketamine IVI
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 6/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=7) | Ketamine SC (N=8) | Ketamine IVI (N=8)
Nausea (General disorders) | 2 (2) | 2 (2) | 4 (4)
Vomiting (General disorders) | 1 (1) | 3 (3) | 1 (1)
Shivering (General disorders) | 3 (3) | 2 (2) | 0 (0)
Sedation (Surgical and medical procedures) | 3 (3) | 1 (1) | 3 (3)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04227704/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT04227704/ICF_001.pdf